CLINICAL TRIAL: NCT03235232
Title: Randomized Clinical Trial to Compare the Efficacy and Safety of BREMEN Eye Drops Versus Combigan in Subjects With Open Angle Glaucoma or Ocular Hypertension
Brief Title: BREMEN Eye Drops Versus Combigan for Open-angle Glaucoma or Intraocular Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: EMS (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EMS0117
Record Dates: First submitted 2017-07-27; First posted 2017-08-01 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Ocular Hypertension; Primary Open-angle Glaucoma
MeSH Terms: conditions — Ocular Hypertension; Glaucoma, Open-Angle | interventions — Brimonidine Tartrate, Timolol Maleate Drug Combination

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BREMEN eye drops (Experimental): 1 drop in affected eye(s), each 12 hours for 8 weeks.
  Interventions: Drug: BREMEN eye drops
- Combigan® (Active Comparator): 1 drop of Combigan® in affected eye(s), each 12 hours for 8 weeks.
  Interventions: Drug: Combigan®

INTERVENTIONS:
Drug: BREMEN eye drops — 1 drop in the affected eye(s), twice a day (approximately each 12 hours) for 8 weeks.
  Arms: BREMEN eye drops
Drug: Combigan® — 1 drop of Combigan® in the affected eye(s), twice a day (approximately each 12 hours) for 8 weeks.
  Arms: Combigan®

SUMMARY:
The purpose of this study is to evaluate the clinical efficacy of the BREMEN eye drops in the treatment of primary open-angle glaucoma or intraocular hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Signed Consent;
* Participants with diagnosis of open-angle glaucoma or hypertension ocular, who needs treatment with drugs association to control the intraocular pressure;
* Participants who have 20/80 visual acuity or more, in both eyes;

Exclusion Criteria:

* Participants with any clinical significant disease that, after evaluation of the investigator, can´t participate in the study;
* Participants with active eye disease, which in the investigator opinion may interfere in the results of this clinical trial;
* Participants presenting previous diagnosis of non-operated cataract, high myopia, high astigmatism, pseudoexfoliation and corneal deformities;
* Participants who had significant visual loss in the last year;
* Treatment-naive participants for open-angle glaucoma or ocular hypertension;
* Participants nonresponders to previous triple combination drug therapy, used in concomitance;
* Participants with previous ocular or intraocular surgery within six months prior to enrollment in the clinical trial;
* Participants with history of hypersensitivity to any formula compounds;
* Participants presenting contraindications to use of beta-adrenergic antagonists;
* Participants diagnosed with uncontrolled cardiovascular disease;
* Participants with severe renal insufficiency or hyperchloremic acidosis;
* Participants in therapy with monoamine oxidase inhibitors (MAOIs);
* Participants who were in use of drugs that can interfere in the evaluation;
* Pregnancy or risk of pregnancy and lactating patients;
* Alcoholism or illicit drug abuse in the last two years;
* Participation in clinical trial in the year prior to this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 406 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
Efficacy based in the reduction of intraocular pressure in patients with open-angle glaucoma or hypertension ocular. | 8 weeks

SECONDARY OUTCOMES:
Safety will be evaluated through the adverse events occurrences | 8 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Allegisa, Campinas, São Paulo, Brazil